CLINICAL TRIAL: NCT05842200
Title: Influence of Selected Lower Limb Biomechanical Variables on Pain, Disability and Balance in Women With Patellofemoral Pain Syndrome: A Cross Sectional Study.
Brief Title: Influence of Selected Lower Limb Biomechanical Variables on Pain, Disability and Balance in Women With PFPS.
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed ElMelhat, Influence of Selected Lower Limb Biomechanical Variables on Pain, Disability and Balance in Women with Patellofemoral Pain Syndrome: A Cross Sectional Study., Cairo University
Other Study IDs: PFPS and lower limb alignment
Record Dates: First submitted 2023-04-24; First posted 2023-05-03 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Patellofemoral Pain Syndrome; Patellofemoral Malalignment Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Device: No

SUMMARY:
Purpose: The aim of this study is to figure out how does the selection of lower-extremity biomechanical variables presented by dynamic knee valgus, tibial torsion and navicular drop may influence pain, disability, and balance in women with patellofemoral pain syndrome.

Methods: Sixty-five women with patellofemoral pain syndrome will be evaluated for lower limb biomechanical variables.

DETAILED DESCRIPTION:
Subjects:

Sixty five women who will be referred by an Orthopedist with patellofemoral pain syndrome diagnosis.

Inclusion criteria:

Women were enrolled in this study according to the following criteria:

1. Female participants with patellofemoral pain syndrome.
2. Age ranges between 18 and 38 years old.
3. Bilateral or unilateral involvement.
4. Minimum score (3 out of 10-point) numerical pain scale (NPR) .
5. Orthopedic clinical confirmation revealing a history of anterior or retro-patellar knee pain aggravated by at least 2 of the following functional activities: 1. prolonged sitting, 2. stairs use, 3. squatting, 4. running, 5. kneeling, 6. hopping/jumping, and/or insidious onset of symptoms unrelated to any traumatic incident and persistent for at least 6 weeks.

Exclusion criteria:

A woman was excluded from the study if she has one or more of the following:

1. History of patellar dislocation or subluxation.
2. Osteoarthritis in the patellofemoral joint.
3. Meniscal or other intraarticular pathologic conditions.
4. cruciate or collateral ligament involvement.
5. Lower limb surgery.
6. Fracture, low back pain condition such as: spondylolisthesis and spondylosis.
7. Neurological deficits.
8. Traumatic injury or any abnormality in the lower extremity.

Methods: Sixty-five women with patellofemoral pain syndrome will be evaluated for dynamic knee valgus using Kinovea software program , tibial torsion using universal goniometer, and navicular drop using calliper.

Numerical pain rating scale (NPRS) will be used to measure pain severity. Arabic version of Kujala score will assess the functional disability in these patients.

Biodex Balance System will screen and will record the Medial-lateral stability index (MLSI), Anterior-posterior stability index (APSI) and an Overall stability index (OSI).

Assessments will be performed in a single session. Then correlation between these variables will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Female participants with patellofemoral pain syndrome.
* Age ranges between 18 and 38 years old.
* Bilateral or unilateral involvement.
* Minimum score (3 out of 10-point) numerical pain scale (NPR)
* Orthopedic clinical confirmation revealing a history of anterior or retro-patellar knee pain aggravated by at least 2 of the following functional activities: 1. prolonged sitting, 2. stairs use, 3. squatting, 4. running, 5. kneeling, 6. hopping/jumping, and/or insidious onset of symptoms unrelated to any traumatic incident and persistent for at least 6 weeks.

Exclusion Criteria:

* History of patellar dislocation or subluxation.
* Osteoarthritis in the patellofemoral joint.
* Meniscal or other intraarticular pathologic conditions.
* Cruciate or collateral ligament involvement.
* Lower limb surgery.
* Fracture, low back pain condition such as: spondylolisthesis and spondylosis.
* Neurological deficits.
* Traumatic injury or any abnormality in the lower extremity

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Sixty-five women with patellofemoral pain syndrome, were included in this study. Individuals were selected from the outpatient clinics present in Cairo University and from private clinics in Cairo and Giza.
  The age of selected women was ranging between 18 and 38 years old. They were able to follow instructions and understand the given commands
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Is there an impact of dynamic knee valgus on pain, disability and balance in women with patellofemoral pain? | baseline
  Dynamic knee valgus is a biomechanical variable that will be measured by Kinovea software program to measure 2D Frontal Plane Projection Angle (2D-FPPA) .
Is there an impact of tibial torsion on pain , disability and balance in women with patellofemoral pain syndrome ? | baseline
  Tibial Torsion will be measured with a universal goniometer with the participant prone on a low table, and with the tested knee bent at 90°.
Is there an impact of navicular drop on pain , disability and balance in women with patellofemoral pain syndrome ? | baseline
  Each participant will be asked to stand barefoot, with weight distributed evenly over each foot. the distance between the navicular tuberosity and the floor will be measured, in millimetres, with a calliper.
Women were assessed using numerical pain rating scale (NPRS) for pain severity. | baseline
  The NPRS has been extensively used to assess pain severity.The Arabic version of NPRS, has been culturally adapted and validated.
Women were assessed by Arabic version of Kujala for functional disability. | baseline
  Kujala Scale, also known as anterior knee pain questionnaire (AKPS), is a self-report tool including 13 knee-specific questions. the Arabic version (AAKPS) has been tested for its validity and reliability in Arabian patients
Women were assessed by Biodex Balance System for balance. | baseline
  Biodex Balance System will screen and will record the Medial-lateral stability index (MLSI), Anterior-posterior stability index (APSI) and an Overall stability index (OSI).

CONTACTS AND LOCATIONS:
Overall Officials: Medhat EM [mmofty], Study Director — Cairo University
Locations (1):
- Ahmed ElMelhat [aelmelhat], Cairo, Egypt

REFERENCES:
- See also: Is spinopelvic sagittal alignment correlated with pain level, functional disability and frontal plane projection angle in women with patellofemoral pain syndrome? A cross-sectional study — https://revistas.um.es/sportk/article/view/537601?fbclid=IwAR3r1CTyCSQKoa-PxlQS207KKTFnNbcXHdighI9mRG-M2Y15XSPf3cUrSVU
- See also: Comparison of selected lower limb biomechanical variables between university of ibadan sportsmen with and without patellofemoral pain syndrome — https://www.sportsmedoa.com/articles/jsmt-aid1046.pdf?fbclid=IwAR3-Ab7YGc6KF_2Jw4TEnBEt_SZ8xjXatNfh5jxuwzBGn6MC8hhHSDHO0qQ